CLINICAL TRIAL: NCT01054300
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, 2-Period, Cross-Over Single Day Evaluation Of The Pharmacokinetic-Pharmacodynamic Effect Of Once And Twice Daily Oral Administration Of PF-04971729 In Patients With Type 2 Diabetes Mellitus
Brief Title: Effects of Once and Twice Daily Dosing Regimen of Ertugliflozin (PF-04971729, MK-8835) In Participants With Type 2 Diabetes (MK-8835-040)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 8835-040; B1521007 (Other: Pfizer Protocol Number); MK-8835-040 (Other: Merck Protocol Number)
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus, Type 2; Adult
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ertugliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Ertu 2 mg/Placebo (Pbo)→Ertu 1 mg/Ertu 1 mg (Experimental): Period 1: Ertu 2 mg in the AM and Pbo in the PM for 1 day. Period 2: Ertu 1 mg in the AM and Ertu 1 mg in the PM for 1 day. There was a >= 7 day washout period between Period 1 and Period 2.
  Interventions: Drug: Ertugliflozin 2 mg single dose; Drug: Ertugliflozin 2 mg split into twice daily; Drug: Placebo
- Cohort 1: Ertu 1 mg/Ertu 1 mg→Ertu 2 mg/Pbo (Experimental): Period 1: Ertu 1 mg in the AM and Ertu 1 mg in the PM for 1 day. Period 2: Ertu 2 mg in the AM and Pbo in the PM for 1 day. There was a >= 7 day washout period between Period 1 and Period 2.
  Interventions: Drug: Ertugliflozin 2 mg single dose; Drug: Ertugliflozin 2 mg split into twice daily; Drug: Placebo
- Cohort 2: Ertu 4 mg/Pbo→Ertu 2 mg/Ertu 2 mg (Experimental): Period 1: Ertu 4 mg in the AM and Pbo in the PM for 1 day. Period 2: Ertu 2 mg in the AM and Ertu 2 mg in the PM for 1 day. There was a >= 7 day washout period between Period 1 and Period 2.
  Interventions: Drug: Ertugliflozin 4 mg single dose; Drug: Ertugliflozin 4 mg split into twice daily; Drug: Placebo
- Cohort 2: Ertu 2 mg/Ertu 2 mg→Ertu 4 mg/Pbo (Experimental): Period 1: Ertu 2 mg in the AM and Ertu 2 mg in the PM for 1 day. Period 2: Ertu 4 mg in the AM and Pbo in the PM for 1 day. There was a >= 7 day washout period between Period 1 and Period 2.
  Interventions: Drug: Ertugliflozin 4 mg single dose; Drug: Ertugliflozin 4 mg split into twice daily; Drug: Placebo

INTERVENTIONS:
Drug: Ertugliflozin 2 mg single dose — Ertugliflozin 2 mg dose (two 1 mg strength tablets), administered as a single dose
  Arms: Cohort 1: Ertu 1 mg/Ertu 1 mg→Ertu 2 mg/Pbo; Cohort 1: Ertu 2 mg/Placebo (Pbo)→Ertu 1 mg/Ertu 1 mg
Drug: Ertugliflozin 2 mg split into twice daily — Ertugliflozin 1 mg dose (1 mg strength tablet) administered twice daily x 1 day
  Arms: Cohort 1: Ertu 1 mg/Ertu 1 mg→Ertu 2 mg/Pbo; Cohort 1: Ertu 2 mg/Placebo (Pbo)→Ertu 1 mg/Ertu 1 mg
Drug: Ertugliflozin 4 mg single dose — Ertugliflozin 4 mg dose (four 1 mg strength tablets), administered as a single dose
  Arms: Cohort 2: Ertu 2 mg/Ertu 2 mg→Ertu 4 mg/Pbo; Cohort 2: Ertu 4 mg/Pbo→Ertu 2 mg/Ertu 2 mg
Drug: Ertugliflozin 4 mg split into twice daily — Ertugliflozin 2 mg dose (two 1 mg strength tablets) administered twice daily x 1 day
  Arms: Cohort 2: Ertu 2 mg/Ertu 2 mg→Ertu 4 mg/Pbo; Cohort 2: Ertu 4 mg/Pbo→Ertu 2 mg/Ertu 2 mg
Drug: Placebo — Placebo to ertugliflozin administered as a single dose

SUMMARY:
This is a Phase 1 randomized, double-blind, sponsor open, 4 arm, 2 way cross-over study using 2 cohorts. The objective of the study is to evaluate the pharmacodynamics (PD) effects and the pharmacokinetic (PK) of single day dosing of 2 mg and 4 mg doses of ertugliflozin (Ertu, PF-04971729/MK-8835) each administered once vs twice daily (morning [AM] and evening [PM]) in adults with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Participants with type 2 diabetes mellitus, either treatment-naïve or on up to 2 acceptable oral anti-diabetes drugs for at least 8-weeks prior to study.

Exclusion Criteria:

* Participants with type 1 diabetes mellitus, participants with stroke, unstable angina, heart attack in last 6-months, uncontrolled blood pressure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-02-17 (Actual); Primary Completion 2010-04-07 (Actual); Study Completion 2010-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Dawra VK, Liang Y, Shi H, Bass A, Hickman A, Terra SG, Zhou S, Cutler D, Sahasrabudhe V. A PK/PD study comparing twice-daily to once-daily dosing regimens of ertugliflozin in healthy subjects . Int J Clin Pharmacol Ther. 2019 Apr;57(4):207-216. doi: 10.5414/CP203343. PMID 30802200
- [Derived] Fediuk DJ, Sahasrabudhe V, Dawra VK, Zhou S, Sweeney K. Population Pharmacokinetic Analyses of Ertugliflozin in Select Ethnic Populations. Clin Pharmacol Drug Dev. 2021 Nov;10(11):1297-1306. doi: 10.1002/cpdd.970. Epub 2021 Jul 2. PMID 34213819

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Ertu 2 mg/Pbo→Ertu 1 mg/Ertu 1 mg: Period 1: Ertugliflozin (Ertu) 2 mg in the AM and placebo (Pbo) in the PM for 1 day. Period 2: Ertu 1 mg in the AM and Ertu 1 mg in the PM for 1 day. There was a >= 7 day washout period between Period 1 and Period 2.
- Cohort 2: Ertu 2 mg/Ertu 2 mg→Ertu 4 mg/P: Period 1: Ertu 2 mg in the AM and Ertu 2 mg in the PM for 1 day. Period 2: Ertu 4 mg in the AM and Pbo in the PM for 1 day. There was a >= 7 day washout period between Period 1 and Period 2.
Period: Period 1
Arm/Group | Cohort 1: Ertu 2 mg/Pbo→Ertu 1 mg/Ertu 1 mg | Cohort 1: Ertu 1 mg/Ertu 1 mg→Ertu 2 mg/Pbo | Cohort 2: Ertu 4 mg/Pbo→Ertu 2 mg/Ertu 2 mg | Cohort 2: Ertu 2 mg/Ertu 2 mg→Ertu 4 mg/P
Started | 13 | 13 | 13 | 13
Completed | 12 (Discontinuation occurred prior to Period 2 dose.) | 13 | 13 | 13
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Period 2
Arm/Group | Cohort 1: Ertu 2 mg/Pbo→Ertu 1 mg/Ertu 1 mg | Cohort 1: Ertu 1 mg/Ertu 1 mg→Ertu 2 mg/Pbo | Cohort 2: Ertu 4 mg/Pbo→Ertu 2 mg/Ertu 2 mg | Cohort 2: Ertu 2 mg/Ertu 2 mg→Ertu 4 mg/P
Started | 12 | 13 | 13 | 13
Completed | 12 | 13 | 12 | 13
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Cohort 1: Period 1: participants received a total daily dose of ertugliflozin 2 mg for 1 day; Period 2: participants received a total daily dose of ertugliflozin 2 mg for 1 day
- Cohort 2: Period 1: participants received a total daily dose of ertugliflozin 4 mg; Period 2: participants received a total daily dose of ertugliflozin 4 mg for 1 day
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Customized [Number; unit: Participants]
  18 - 44 years | 7 | 7 | 14
  45 - 64 years | 17 | 18 | 35
  65 years or older | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Urinary Glucose Excretion Over 0 to 24 Hours
Description: Urine for analysis of glucose was collected at prespecified intervals. Each participant emptied his/her bladder just before dosing, and the collection started after the morning dose (collection times: 0-4 hours, 4-8 hours, 8-12 hours, and 12-24 hours after the morning dose). The average amount of urinary glucose excreted from 0 to 24 hours after the morning dose is presented in the table below.
Time Frame: 0 to 24 hours after the morning dose
Population: Analysis population included randomized participants who received assigned dose and had urine collection during all of the collection time frames between 0 and 24 hours following the morning dose.
Measure: Least Squares Mean (90% Confidence Interval); unit: Grams
Groups:
- Cohort 1: Ertugliflozin 1 mg Twice Daily: Participants received ertugliflozin 1 mg twice daily for 1 day
- Cohort 1: Ertugliflozin 2 mg Once Daily: Participants received ertugliflozin 2 mg once daily for 1 day
- Cohort 2: Ertugliflozin 2 mg Twice Daily: Participants received ertugliflozin 2 mg twice daily for 1 day
- Cohort 2: Ertugliflozin 4 mg Once Daily: Participants received ertugliflozin 4 mg once daily for 1 day
Arm/Group | Cohort 1: Ertugliflozin 1 mg Twice Daily | Cohort 1: Ertugliflozin 2 mg Once Daily | Cohort 2: Ertugliflozin 2 mg Twice Daily | Cohort 2: Ertugliflozin 4 mg Once Daily
Number analyzed (Participants) | 25 | 25 | 24 | 24
Grams | 69.45 (9.08) [54.20 to 84.70] | 70.43 (9.08) [55.19 to 85.68] | 78.29 (9.77) [61.87 to 94.72] | 80.54 (9.81) [64.05 to 97.02]

2. Primary Outcome: Urinary Glucose Excretion by Time Period
Description: Urine for analysis of glucose was collected at prespecified intervals. Each participant emptied his/her bladder just before dosing, and the collection started after the morning dose (collection times: 0-4 hours, 4-8 hours, 8-12 hours, and 12-24 hours after the morning dose). The average amount of urinary glucose excreted during the pre-specified time frame is presented in the table below.
Time Frame: At 0-4 hrs, 4-8 hrs, 8-12 hrs, and 12-24 hrs after the AM dose (up to 24 hours)
Population: Analysis population included randomized participants who received assigned dose and had urine collection during the specific time frame.
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Cohort 1: Ertugliflozin 1 mg Twice Daily | Cohort 1: Ertugliflozin 2 mg Once Daily | Cohort 2: Ertugliflozin 2 mg Twice Daily | Cohort 2: Ertugliflozin 4 mg Once Daily
Number analyzed (Participants) | 25 | 26 | 25 | 26
Grams
  0 to 4 hours post dose | 12.88 (14.66) | 14.03 (11.63) | 14.66 (11.81) | 16.34 (10.16)
  4 to 8 hours post dose: number analyzed (Participants) | 25 | 25 | 25 | 25
  4 to 8 hours post dose | 15.42 (12.00) | 17.87 (12.60) | 16.97 (11.64) | 19.78 (14.02)
  8 to 12 hours post dose: number analyzed (Participants) | 25 | 26 | 24 | 25
  8 to 12 hours post dose | 14.47 (8.84) | 11.99 (7.70) | 14.30 (10.52) | 12.91 (6.93)
  12 to 24 hours post dose: number analyzed (Participants) | 25 | 26 | 24 | 26
  12 to 24 hours post dose | 26.76 (20.10) | 26.31 (21.11) | 31.47 (22.71) | 32.94 (21.08)

3. Primary Outcome: 24-hour Weighted Mean Plasma Glucose
Description: Blood was collected during each treatment period at pre-dose (fasted) on Day 1 (Hour 0) and post-dose (fed) on Day 1 at 0.5, 1, 2, 3, 4, 5, 5.5, 6, 7, 8, 10, 12, 12.5, 13, 14, 15, 16, 18, and 24 hours.
Time Frame: Up to 24 hours
Population: Analysis population included randomized participants who received study drug and had mean plasma glucose measurements during all of the specific collection time frames.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cohort 1: Ertugliflozin 1 mg Twice Daily | Cohort 1: Ertugliflozin 2 mg Once Daily | Cohort 2: Ertugliflozin 2 mg Twice Daily | Cohort 2: Ertugliflozin 4 mg Once Daily
Number analyzed (Participants) | 23 | 25 | 23 | 24
mg/dL | 173.6 (26.94) | 175.7 (29.88) | 169.1 (35.91) | 170.4 (41.26)

4. Primary Outcome: Weighted Mean Postprandial Plasma Glucose
Description: The weighted mean postprandial glucose over the specified intervals were analyzed by cohort.
Time Frame: At 0-5 hours, 5-12 hrs, and 12-18 hrs after the morning dose (up to 18 hours)
Population: Analysis population included randomized participants who received assigned dose and had postprandial plasma glucose measurements during the specific time frame.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cohort 1: Ertugliflozin 1 mg Twice Daily | Cohort 1: Ertugliflozin 2 mg Once Daily | Cohort 2: Ertugliflozin 2 mg Twice Daily | Cohort 2: Ertugliflozin 4 mg Once Daily
Number analyzed (Participants) | 25 | 26 | 25 | 25
mg/dL
  0 to 5 hours | 200.1 (38.27) | 187.2 (41.37) | 194.1 (46.87) | 189.9 (53.17)
  5 to 12 hours | 159.4 (25.76) | 159.8 (28.46) | 160.5 (42.14) | 161.5 (40.70)
  12 to 18 hours: number analyzed (Participants) | 25 | 26 | 24 | 25
  12 to 18 hours | 180.7 (35.98) | 190.7 (35.38) | 182.6 (40.79) | 181.9 (40.79)

5. Primary Outcome: Fasting Plasma Glucose
Description: Blood samples were to be collected following a fast from all food and drink (except water) for at least 8 hours. Fasting Plasma Glucose was collected as part of the assessment of weighted mean 24-hour plasma glucose. As such, it was not specified as an endpoint in the Statistical Analysis Plan and was not analyzed or summarized separately.
Time Frame: Up to 24 hours
Population: The protocol listed fasting plasma glucose as one of the endpoints of the study. However, given the assessment of weighted mean 24-hour plasma glucose and weighted mean postprandial glucose following the 3 meals on Day 1 of each period, analysis of fasting plasma glucose was not undertaken.
Arm/Group | Cohort 1: Ertugliflozin 1 mg Twice Daily | Cohort 1: Ertugliflozin 2 mg Once Daily | Cohort 2: Ertugliflozin 2 mg Twice Daily | Cohort 2: Ertugliflozin 4 mg Once Daily
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Primary Outcome: Fasting C-peptide
Description: The fasting c-peptide was analyzed by cohort using a mixed-effects model with sequence, period, and treatment as fixed effects and participant within sequence as a random effect.
Time Frame: Up to 24 hours (0 and 24 hours)
Population: Analysis population included randomized participants who received assigned dose and had fasting c-peptide measurements during the specific time frame.
Measure: Least Squares Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Cohort 1: Ertugliflozin 1 mg Twice Daily | Cohort 1: Ertugliflozin 2 mg Once Daily | Cohort 2: Ertugliflozin 2 mg Twice Daily | Cohort 2: Ertugliflozin 4 mg Once Daily
Number analyzed (Participants) | 25 | 26 | 25 | 26
ng/mL | 2.82 (1.148) [2.54 to 3.11] | 2.76 (0.997) [2.47 to 3.04] | 3.00 (0.916) [2.64 to 3.35] | 2.99 (0.973) [2.64 to 3.34]

7. Primary Outcome: Number of Participants Experiencing an Adverse Event
Description: An adverse event is any untoward medical occurrence in a clinical investigation participant administered a product or medical device. The table below includes all data collected since the first dose of study drug.
Time Frame: Up to 16 days
Population: Analysis population includes all treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ertugliflozin 1 mg Twice Daily | Cohort 1: Ertugliflozin 2 mg Once Daily | Cohort 2: Ertugliflozin 2 mg Twice Daily | Cohort 2: Ertugliflozin 4 mg Once Daily
Number analyzed (Participants) | 25 | 26 | 26 | 26
Participants | 5 | 8 | 3 | 5

8. Primary Outcome: Number of Participants Discontinuing Study Drug Due to an Adverse Event
Description: An adverse event is any untoward medical occurrence in a clinical investigation participant administered a product or medical device. The table below includes all data collected since the first dose of study drug. Data include participants discontinued due to adverse events, participants with dose reduced or temporary discontinuation due to adverse events.
Time Frame: Up to 8 days (Day 1 in each dosing period)
Population: Analysis population includes all treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Ertugliflozin 1 mg Twice Daily | Cohort 1: Ertugliflozin 2 mg Once Daily | Cohort 2: Ertugliflozin 2 mg Twice Daily | Cohort 2: Ertugliflozin 4 mg Once Daily
Number analyzed (Participants) | 25 | 26 | 26 | 26
Participants | 0 | 1 | 0 | 0

9. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time 0 to Time of the Last Quantifiable Concentration (AUClast) for Ertugliflozin
Description: Pharmacokinetic (PK) parameter of AUClast for study drug. Actual sample collection times (relative to the AM dose) were used for the pharmacokinetic analysis.
Time Frame: 0 predose, 0.5, 1, 2, 3, 4, 5, 5.5, 6, 7, 8, 10, 12, 18, 24 hours postdose
Population: All participants randomized and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1: Ertugliflozin 1 mg Twice Daily | Cohort 1: Ertugliflozin 2 mg Once Daily | Cohort 2: Ertugliflozin 2 mg Twice Daily | Cohort 2: Ertugliflozin 4 mg Once Daily
Number analyzed (Participants) | 25 | 26 | 25 | 26
ng*hr/mL | 131.8 (26) | 132.7 (28) | 272 (19) | 270.5 (20)

10. Primary Outcome: Maximum Plasma Concentration (Cmax) of Ertugliflozin
Description: PK parameter of Cmax for study drug. Actual sample collection times (relative to the AM dose) were used for the pharmacokinetic analysis.
Time Frame: 0 predose, 0.5, 1, 2, 3, 4, 5, 5.5, 6, 7, 8, 10, 12, 18, 24 hours postdose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: Ertugliflozin 1 mg Twice Daily | Cohort 1: Ertugliflozin 2 mg Once Daily | Cohort 2: Ertugliflozin 2 mg Twice Daily | Cohort 2: Ertugliflozin 4 mg Once Daily
Number analyzed (Participants) | 25 | 26 | 25 | 26
ng/mL | 19.51 (39) | 26.98 (37) | 34.80 (23) | 50.83 (25)

11. Primary Outcome: Time Taken to Reach the Maximum Observed Plasma Concentration (Tmax) of Ertugliflozin
Description: PK parameter of Tmax for study drug. Actual sample collection times (relative to the AM dose) were used for the pharmacokinetic analysis.
Time Frame: 0 predose, 0.5, 1, 2, 3, 4, 5, 5.5, 6, 7, 8, 10, 12, 18, 24 hours postdose
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: Ertugliflozin 1 mg Twice Daily | Cohort 1: Ertugliflozin 2 mg Once Daily | Cohort 2: Ertugliflozin 2 mg Twice Daily | Cohort 2: Ertugliflozin 4 mg Once Daily
Number analyzed (Participants) | 25 | 26 | 25 | 26
hours | 6.00 [0.500 to 12.0] | 1.00 [0.500 to 5.50] | 6.00 [0.500 to 8.00] | 1.00 [0.500 to 6.00]

ADVERSE EVENTS:
Time Frame: Up to 16 days (including 7-day follow-up for each period)
Arm/Group | Cohort 1: Ertugliflozin 1 mg Twice Daily | Cohort 1: Ertugliflozin 2 mg Once Daily | Cohort 2: Ertugliflozin 2 mg Twice Daily | Cohort 2: Ertugliflozin 4 mg Once Daily
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 5/25 | 8/26 | 3/26 | 5/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Ertugliflozin 1 mg Twice Daily (N=25) | Cohort 1: Ertugliflozin 2 mg Once Daily (N=26) | Cohort 2: Ertugliflozin 2 mg Twice Daily (N=26) | Cohort 2: Ertugliflozin 4 mg Once Daily (N=26)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomitting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 1 (1) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution will provide manuscripts, abstracts, or the full text of any other intended disclosure (poster presentation, invited speaker or guest lecturer presentation, etc.) to Pfizer at least 30 days before they are submitted for publication or otherwise disclosed. If any patent action is required to protect intellectual property rights, Institution agrees to delay the disclosure for a period not to exceed an additional 60 days.